CLINICAL TRIAL: NCT00286520
Title: Treatment of Fecal Incontinence and Constipation in Patients With Spinal Cord Injury - a Prospective, Randomized, Controlled, Multicentre Trial of Transanal Irrigation Vs. Conservative Bowel Management
Brief Title: Treatment of Fecal Incontinence and Constipation in Patients With Spinal Cord Injury
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Coloplast A/S (Industry); Montecatone Rehabilitation Institute S.p.A. (Other); National Spinal Injuries Centre, Stoke Mandeville Hospital, United Kingdom, (Unknown); Orthopädische Universitätsklinik Heidelberg, Germany, (Unknown); Karolinska University Hospital (Other); Central Jutland Regional Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DK021CC
Record Dates: First submitted 2006-01-30; First posted 2006-02-03 (Estimated); Last update posted 2006-02-03 (Estimated); Status verified 2006-02

CONDITIONS: Constipation; Fecal Incontinence; Spinal Cord Injury
Keywords: Constipation; Fecal incontinence; Spinal cord injury; transanal irrigation; quality of life
MeSH Terms: conditions — Constipation; Fecal Incontinence; Spinal Cord Injuries

INTERVENTIONS:
Procedure: Transanal irrigation with Peristeen Anal Irrigation

SUMMARY:
The study aims to compare a newly developed system for transanal colonic irrigation (Peristeen Anal Irrigation) with a bowel management regime that does not include irrigation in a prospective, randomized trial in spinal cord lesion patients (SCL- patients) with faecal incontinence and/or constipation.

Population; 80 SCL- patients with faecal incontinence and/or constipation from five countries.

Focus on:

Bowel symptom score Neurogenic Bowel Dysfunction score Symptom related quality of life questionnaire Time expenditure for performance of bowel care ans side effects

DETAILED DESCRIPTION:
The magnitude of bowel dysfunction in spinal cord injury patients has been documented in several studies. Spinal cord injury affects colorectal motility, transit times, and bowel emptying often leading to constipation, fecal incontinence or a combination of both. Although these symptoms are not life-threatening, they may have a severe impact on quality of life as well as increase levels of anxiety and depression.

Various bowel management programs have been empirical, and individual solutions have been sought on a trial-and-error basis. Transanal irrigation has been used in selected patients with constipation or fecal incontinence. The majority of spinal cord injured patients in a recent study benefited from the treatment. However, there is limited evidence in the literature supporting any bowel management program in spinal cord injury in favor of another and well-designed controlled trials are still lacking. Therefore, the present study aims to compare transanal irrigation with conservative bowel management, defined as best supportive bowel care without irrigation, in a prospective, randomized, controlled, multicentre study among spinal cord injured patients with neurogenic bowel dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over
* Spinal cord lesion at any level at least 3 months from injury
* At least one or more of the following symptoms:
* Spending ½ hour or more attempting to defecate each day or every second day
* Symptoms of autonomic dysreflexia before or during defecation
* Abdominal discomfort before or during defecation
* Episodes of faecal incontinence once or more per month
* The patient is able to understand the treatment and is willing to comply with the prescribed regimen
* The patient is able to perform transanal colonic irrigation seated on a toilet commode with or without assistance
* Signed informed consent has been obtained

Exclusion Criteria:

* Co-existing major unsolved physical problems due to the injury
* Perform transanal retrograde irrigation on a regular basis
* Evidence of bowel obstruction
* Evidence of inflammatory bowel disease
* History of cerebral palsy or cerebral apoplexy
* Multiple sclerosis
* Diabetic polyneuropathy
* Previous abdominal or perianal surgery (not including minor surgery as appendectomy or haemorrhoidectomy)
* Pregnant or lactating
* Evidence of spinal chock
* Mentally unstable
* Treatment with more than 5 mg prednisolon per day.
* PNS implant (sacral nerve stimulation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2003-12; Study Completion 2005-08

PRIMARY OUTCOMES:
Cleveland Clinic Constipaton Scoring System
St. Mark's Fecal Incontinence Grading System

SECONDARY OUTCOMES:
Neurogenic Bowel Dysfunction Score
American Society of Colorectal Surgeon Fecal Incontinence Score

CONTACTS AND LOCATIONS:
Overall Officials: Soeren Laurberg, professor, D.M.Sci, Study Chair — Surgical Research Unit, Department of Surgery P, Aarhus University Hospital, Denmark
Locations (1):
- Surgical Research Unit, Department of Surgery P, Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Background] Christensen P, Olsen N, Krogh K, Bacher T, Laurberg S. Scintigraphic assessment of retrograde colonic washout in fecal incontinence and constipation. Dis Colon Rectum. 2003 Jan;46(1):68-76. doi: 10.1007/s10350-004-6498-0. PMID 12544524
- [Background] Christensen P, Kvitzau B, Krogh K, Buntzen S, Laurberg S. Neurogenic colorectal dysfunction - use of new antegrade and retrograde colonic wash-out methods. Spinal Cord. 2000 Apr;38(4):255-61. doi: 10.1038/sj.sc.3100991. PMID 10822397
- [Background] Krogh K, Olsen N, Christensen P, Madsen JL, Laurberg S. Colorectal transport during defecation in patients with lesions of the sacral spinal cord. Neurogastroenterol Motil. 2003 Feb;15(1):25-31. doi: 10.1046/j.1365-2982.2003.00381.x. PMID 12588466